CLINICAL TRIAL: NCT00736970
Title: A Phase II Trial of Oral Deforolimus (AP23573; MK-8669), an mTOR Inhibitor, in Combination With Trastuzumab for Patients With HER2-positive Trastuzumab-Refractory Metastatic Breast Cancer
Brief Title: Oral Deforolimus With Trastuzumab for Patients With HER2-positive Trastuzumab-Refractory Metastatic Breast Cancer (8669-009)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-009; AP23573-08-207 (Other: Secondary ID)
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: ridaforolimus; deforolimus; AP23573; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ridaforolimus; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 10 mg oral tablets administered at 40 mg once daily for 5 consecutive days each week, followed by 2 days without ridaforolimus
  Interventions: Drug: ridaforolimus; Drug: trastuzumab

INTERVENTIONS:
Drug: ridaforolimus — 10 mg oral tablets administered at 40 mg once daily for 5 consecutive days each week, followed by 2 days without ridaforolimus.
  Other Names: deforolimus; AP23573; MK-8669; ridaforolimus was also known as deforolimus until May 2009
Drug: trastuzumab — single intravenous infusion every week; initial dose of 4 mg/kg over 90 minutes, then 2 mg/kg over 30 minutes
  Other Names: Herceptin

SUMMARY:
This clinical trial will study the use of ridaforolimus in metastatic breast cancer subjects whose tumors have shown a resistance to trastuzumab (herceptin). The goal of this study is to find out if subjects treated with ridaforolimus in combination with trastuzumab have a positive response to the treatment, and if treatment with ridaforolimus in combination with trastuzumab prolongs survival.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 years of age or older
* Histologically confirmed HER2-positive metastatic breast cancer
* Trastuzumab-resistance
* Measurable disease, according to RECIST guidelines
* ECOG performance status less than or equal to 1
* Life expectancy greater than 3 months
* No prior treatment with temsirolimus, everolimus, rapamycin, or any other mTOR inhibitor
* At least 4 weeks must have lapsed between prior investigational therapy, chemotherapy or radiotherapy, and the first dose of ridaforolimus
* Left ventricular ejection greater than or equal to 50%
* Adequate cardiovascular function
* Adequate hematological, hepatic, and renal function
* Serum cholesterol less than or equal to 350 mg/dL and triglycerides less than or equal to 400 mg/dL
* Negative pregnancy test within 7 days prior to first dose of study drug and must use an approved contraceptive method from screening to 30 days after the last dose of study drug
* Availability and patient consent to obtain archival tissue samples
* Signed informed consent

Exclusion Criteria:

* Inadequate recovery from any prior surgical procedure or having undergone any major surgery within 2 weeks before trial entry
* Grade 1 or Grade 2 hypersensitivity reactions to prior trastuzumab therapy if these reactions prevented further trastuzumab administration
* Grade 3 or Grade 4 hypersensitivity reaction to prior trastuzumab
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs, resulting in dyspnea at rest
* Known allergy to macrolide antibiotics
* Pregnant or breast-feeding
* Know history of HIV
* Diagnosis of brain metastasis or leptomeningeal carcinomatosis within 3 months
* Other malignancies within the past 3 years, except for adequately treated carcinoma of the cervix or basal or squamous cell carcinoma of the skin
* Active infection requiring prescription intervention
* Newly diagnosed or poorly controlled Type 1 or 2 diabetes
* Other concurrent illness which, in the Investigator's judgment, would either compromise the patient's safety or interfere with the evaluation of the safety of the study drug
* Concurrent treatment with medications that strongly induce or inhibit cytochrome P450.
* Any condition that renders patient unable to fully understand and provide informed consent and/or comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-07; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) measured by modified RECIST guidelines | Duration of the study

SECONDARY OUTCOMES:
Characterize the overall safety and tolerability of oral deforolimus administered in combination with standard dose trastuzumab | Duration of the study
Evaluate the clinical-benefit response rate (CR or PR, or SD ≥ six 4-week cycles) | Throughout the trial
Evaluate additional efficacy endpoints, such as duration of response, time to tumor progression, progression-free survival, progression free survival rate, and overall survival | Duration of the trial
Perform exploratory molecular analyses | Duration of the trial

REFERENCES:
- [Result] Seiler M, Ray-Coquard I, Melichar B, Yardley DA, Wang RX, Dodion PF, Lee MA. Oral ridaforolimus plus trastuzumab for patients with HER2+ trastuzumab-refractory metastatic breast cancer. Clin Breast Cancer. 2015 Feb;15(1):60-5. doi: 10.1016/j.clbc.2014.07.008. Epub 2014 Aug 17. PMID 25239224